CLINICAL TRIAL: NCT04910698
Title: Efficacy of Antibiotic Short Course for Bloodstream Infections in Acute Myeloid Leukemia Patients With Febrile Neutropenia: a Retrospective Comparative Study
Brief Title: Efficacy of Antibiotic Short Course for Bloodstream Infections in Acute Myeloid Leukemia Patients With Febrile Neutropenia
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Antibioshort neutropenia
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Bloodstream Infection; Acute Myeloid Leukemia; Febrile Neutropenia
Keywords: antibiotic short course, appropriate use of antibiotics
MeSH Terms: conditions — Sepsis; Leukemia, Myeloid, Acute; Febrile Neutropenia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short course treatment: Patients who received antibiotic for 7 or less days, except for nonfermenting bacteria and Staphylococcus aureus or lugdunensis for which the threshold was 10 days and 14 days, respectively.
  Interventions: Drug: Antibiotic
- Long course treatment: Patients who received antibiotic for more than 7 days, except for nonfermenting bacteria and Staphylococcus aureus or lugdunensis for which the threshold was 10 days and 14 days, respectively.
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Antibiotic duration of treatment defined if the patient belonged to long course or short course group.

SUMMARY:
There is no specific recommendation about antimicrobial treatment length for documented infections in chemotherapy induced febrile neutropenia. The aim of this study was to compare long versus short antibiotic course for bloodstream infection treatment in acute myeloid leukemia patients during febrile neutropenia. This monocentric retrospective comparative study included all consecutive bloodstream infection episodes among acute myeloid leukemia patients with febrile neutropenia for 3 years (2017-2019). Episodes were classified regarding the length of antibiotic treatment, considered as short course if the treatment lasted ≤7 days, except for nonfermenting bacteria and Staphylococcus aureus or lugdunensis for which the threshold was ≤10 days and ≤14 days, respectively. The primary outcome was the number of bloodstream infection relapses in both groups within 30 days of antibiotic discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia
* chemo-induced febrile neutropenia
* Bloodstream infection

Exclusion Criteria:

* lack of data
* endovascular infections
* surgical treatment required
* central nervous system infections
* antibiotic treatment < 4 days
* death before the end of antibiotic treatment
* unappropriated antibiotic treatment at 48h
* relapses of bloodstream infection episodes already included
* hematopoietic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All bloodstream infection episodes occuring in patients suffering from febrile neutropenia during acute myeloid leukemia between January 2017 and December 2019 in University Hospital of Poitiers were included.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Bloodstream infection relapses | within 30 days of antibiotic discontinuation
  The primary outcome was to compare the number of bloodstream infection relapses in both groups within 30 days of antibiotic discontinuation.

SECONDARY OUTCOMES:
Mortality | within 30 days of antibiotic discontinuation
  Comparison of mortality rate within 30 days of antibiotic discontinuation
Epidemiology of bacteria | at baseline
  Distribution of bacteria responsible for bloodstream infection
Risk factors for relapses | within 30 days of antibiotic discontinuation
  Analyse of risk factors for bloodstream infection relapses

CONTACTS AND LOCATIONS:
Overall Officials: France Cazenave-Roblot, Study Director
Locations (1):
- University Hospital, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided